CLINICAL TRIAL: NCT06872177
Title: Axial Inclination of Mandibular Molar Dental Implants Versus Natural Teeth: What Are the Differences?
Brief Title: Chart Review: Comparing the Position and Tilt of Dental Implants Versus Those of Natural Teeth
Status: Not yet recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Binnaz Leblebicioglu, Professor, Ohio State University
Other Study IDs: 2025H0006
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dental Implant
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chart Review: Existing records of patients at the Ohio State University College of Dentistry who had a dental implant of one single molar tooth between January 1, 2016 and January 6, 2025
  Interventions: Other: Measurements

INTERVENTIONS:
Other: Measurements — On existing identified chart records: measurements on CBCT and panographic radiographs.

SUMMARY:
Background:

When placing a dental implant, it is not always possible to place it exactly in the same position as the tooth that it replaced. That might be because of how the gums and mouth are shaped, since some bone is always lost after a tooth is extracted. Researchers want to study the records of people who have had dental implants. They want to check to see how much difference there is between how the implant is positioned and how the same tooth on the other side is positioned. They also want to compare how the implant is positioned compared to the tooth it replaced, when that is possible in the dental record.

Study design:

This study will not enroll any participants. The researchers will search the database of patient records at the study clinic to find people who have had dental implants of a single molar tooth. Then they will look at them to find records that include good images that they can use to compare the implant and tooth positions.

Researchers will then analyze the findings and write a review article.

DETAILED DESCRIPTION:
This is a retrospective chart review. Specifically, the clinic e-chart system will be used to locate patients who received implant surgery. E-charts from January 1, 2016, to January 6, 2025, with pre- and post-implant surgery tomography (CBCT) documentation will be identified and used for this study.

Demographic and clinical data (age, sex, systemic conditions, implant details and surgical treatment outcomes) related to these cases will be collected. Radiographic measurements will include the following:

* On tomography: 1. Buccolingual axial inclination of natural molars and implants. 2. Mesiodistal axial inclination of natural molars and implants. 3. Presence/absence of fenestration and/or dehiscence around implants 4. Proximity to mandibular canal and/or foramen mentale
* On Panoramic radiograph: Mesiodistal axial inclination of natural molars and implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular molar implant placement.
* Presence of contralateral natural mandibular first, second molars or both.
* Availability of pre-extraction CBCT scans of the corresponding or contralateral mandibular molar tooth or panoramic radiographs for mesiodistal angulation.
* Availability of post-implant CBCT scans or panoramic radiographs for mesiodistal angulation

Exclusion Criteria:

* Incomplete or low-quality CBCT scans.
* History of mandibular trauma or pathologies altering tooth or implant alignment.
* History of reconstructive mandibular surgery in the implant region.
* History of periapical pathology

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing records of patients at the Ohio State University College of Dentistry who have had a dental implant of one single molar tooth, between January 1, 2016 and January 6, 2025
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Replaced Tooth Comparison | Baseline (prior to tooth extraction), day 1 of implant placement, day 1 of crown placement (4-6 months after implant placement)
  Difference in buccolingual and mesiodistal angulations of placed implant compared with pre-extraction natural tooth.
Contralateral Tooth Comparison | Day 1 of implant placement, day 1 of crown placement (4-6 months after implant placement)
  Difference in buccolingual and mesiodistal angulations of placed implant compared with contralateral natural molar.

OTHER OUTCOMES:
Frequency of Fenestration/Dehiscence | Day 1 of crown placement (4-6 months post-implant placement)
  Presence/absence of fenestration and/or dehiscence around implants
Distance from Foramen Mentale | Day 1 of crown placement (4-6 months post-implant placement)
  Distance between the implant and the foramen mentale, measured with software on CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Binnaz Leblebicioglu, DDS, MMS, PhD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No